CLINICAL TRIAL: NCT05177302
Title: Restoration of Lumbopelvic Movement Control: Effect of Injury History, and the Role of Cortical Control and Its Practical Application(3)
Brief Title: Lumbopelvic Movement Control: Effect of Injury History, and the Role of Cortical Control and Its Practical Application 3
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Other Study IDs: YM110027E(3)
Record Dates: First submitted 2021-12-02; First posted 2022-01-04 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Patient Reported Outcome
Keywords: hip and/ or groin pain; reliability; validity; responsiveness; HAGOS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with hip and/ or groin pain: The young to middle-aged physically active individuals with hip and/ or groin pain, which symptoms lasting for 2 to 6 month.
  Interventions: Other: HAGOS-C; Other: SF-36v2

INTERVENTIONS:
Other: HAGOS-C — The subjects will be instructed to complete HAGOS-C at the initial contact and again after 1 week and 4 month for reliability and responsiveness test, respectively
Other: SF-36v2 — The subjects will be instructed to complete SF-36v2 at the initial contact to determine the validity of HAGOS-C

SUMMARY:
Hip and groin pain is a common injury in athletes participating multidirectional sports, and resulting in decreased sports participation and quality of life. The Copenhagen Hip And Groin Outcome Score (HAGOS) specifically targets young to middle-aged physically active individuals with long-standing hip and/ or groin pain, it consists of six separate subscales about symptoms, pain, physical function in daily living, physical function in sports and recreation, participation in physical activities and hip and/ or groin related quality of life (QoL), which all subscales have shown to have adequate validity, reliability and responsiveness in the original version of the questionnaire. Lacking of the specifical questionnaire for physically active people with hip and/or groin pain, the purpose of the study is to translate and cross-culturally adapt HAGOS into Chinese version (HAGOS-C) according to the guidelines from Beaton et al.

DETAILED DESCRIPTION:
Hip and groin pain is a common injury in athletes participating multidirectional sports, and resulting in decreased sports participation and quality of life. The Copenhagen Hip And Groin Outcome Score (HAGOS) specifically targets young to middle-aged physically active individuals with long-standing hip and/ or groin pain, it consists of six separate subscales about symptoms, pain, physical function in daily living, physical function in sports and recreation, participation in physical activities and hip and/ or groin related quality of life (QoL), which all subscales have shown to have adequate validity, reliability and responsiveness in the original version of the questionnaire. Lacking of the specifical questionnaire for physically active people with hip and/or groin pain, the purpose of the study is to translate and cross-culturally adapt HAGOS into Chinese version (HAGOS-C) according to the guidelines from Beaton et al.

We translated the questionnaire from the English version involved following steps: (1)initial translation with two bilingual translators (2) holding consensus meeting for the preliminary Chinese version (3) back translation with other two bilingual back translators (4) another consensus meeting for ensuring the consistency with original English version (5) pretesting for wording and understanding (6) Wording, rephrasing and format corrected to obtain final Chinese version of the HAGOS.

The aim of the study is to determine the validity, reliability and responsiveness of HAGOS-C by recruiting young to middle-aged physically active individuals with long-standing hip and/ or groin pain.

ELIGIBILITY:
Inclusion Criteria:

* physically active at least 2.5 hrs/week
* tenderness on iliopsoas, inguinal, hip adductors, pubic symphysis
* hip and/ or groin pain during motion with restriction or giving way sensation, or clicking sound in hip joint.
* pain lasting for 2 to 6 month and no obvious changes within 3 week recently.

Exclusion Criteria:

* other symptoms in lumbar, knee or ankle joint.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The individuals with long-standing hip and/ or groin pain lasting 2 to 6 month, which hip and/ or groin pain during motion with restriction or giving way sensation, or clicking sound in hip joint, and tenderness on iliopsoas, inguinal, hip adductors, pubic symphysis will be included . The individuals with other symptoms in lumbar, knee or ankle joint will be excluded.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
HAGOS-C | immediately after the intervention
  The individuals will be asked to complete 37 items of the HAGOS-C after instruction
SF-36v2 | immediately after the intervention
  The individuals will be asked to complete 36 items of the SF-36v2 after instruction for validation
HAGOS-C | after 1 week
  The individuals will be asked to complete 37 items of the HAGOS-C after instruction for reliability.
HAGOS-C | after 4 months
  The individuals will be asked to complete 37 items of the HAGOS-C after instruction for responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fen Shih, Ph.D, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming Chiao-Tung University
Locations (1):
- National Yang Ming University, Taipei, Taiwan